CLINICAL TRIAL: NCT05449184
Title: A Prospective, Randomized, Controlled Clinical Study of Balloon Eustachian Tuboplasty Combined With Tympanostomy Tube Insertion in the Treatment of Intractable Otitis Media With Effusion After Radiotherapy for Nasopharyngeal Carcinoma
Brief Title: A Prospective, Randomized, Controlled Clinical Study of BET Combined With Tympanostomy Tube Insertion in the Treatment of Intractable OME After Radiotherapy for NPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-123
Record Dates: First submitted 2022-06-01; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-05

CONDITIONS: Otitis Media With Effusion After Nasopharyngeal Carcinoma
Keywords: Balloon Eustachian Tuboplasty; Tympanostomy Tube Insertion; Otitis Media With Effusion; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Otitis Media with Effusion; Nasopharyngeal Carcinoma | interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon Eustachian Tuboplasty with Tympanostomy Tube Insertion (Experimental)
  Interventions: Procedure: Balloon Eustachian Tuboplasty with Tympanostomy Tube Insertion
- Tympanostomy Tube Insertion (Other)
  Interventions: Procedure: Tympanostomy Tube Insertion

INTERVENTIONS:
Procedure: Balloon Eustachian Tuboplasty with Tympanostomy Tube Insertion — Under local or general anesthesia, insert a balloon into one Eaustachian tube and inflate it for up to two minutes. The balloon is then removed. Subsequently, pierce the tympanic membrane in the front and lower quadrants, suck the tympanic effusion, and then insert a tympanic ventilation tube. The tube will be removed 6 months later.
  Arms: Balloon Eustachian Tuboplasty with Tympanostomy Tube Insertion
Procedure: Tympanostomy Tube Insertion — Under local or general anesthesia, pierce the tympanic membrane in the front and lower quadrants, suck the tympanic effusion, and then insert a tympanic ventilation tube. The tube will be removed 6 months later.
  Arms: Tympanostomy Tube Insertion

SUMMARY:
The primary purpose of this study is to compare balloon Eustachian tuboplasty (BET) combined with tympanostomy tube insertion and simply tympanostomy tube insertion in the treatment of otitis media with effusion (OME) in post-radiotherapy patients on the improvement of subjective symptoms (ear fullness, etc.) and the tympanogram.

The secondary purpose is to clarify the effects of BET on the incidence of middle ear infection and slippage of ventilation tube during tube retention, as well as to determine the difference of hearing improvement between the two management methods.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is the most common malignancy of the nasopharynx, of which Guangdong Province is the high-risk area. At present, the comprehensive treatment plan based on radiotherapy (RT) makes NPC a good prognosis, so it is the complications of RT that have become the main factor affecting the life quality of patients. Otitis media with effusion (OME) following RT is the most common ear complication, which is characterized by a large amount of effusion from the tympanic cavity (the cavity of middle ear).

Ear fullness and hearing loss could take place because of tympanic effusions, reducing the patient's ability to communicate and increasing life risk. Currently Eustachian tube dysfunction (ETD) due to RT is regarded as an important causative factor.

The Eustachian tube, connecting the middle ear to the outside world, is an important ventilation pipe. RT could lead to hyperemia, edema, and then fibrosis and atrophy of the Eustachian tube mucosa, resulting in organic changes of the Eustachian tube, including stiffness, adhesions, narrowing and even atresia, and eventually the formation of OME.

Comparatively, non-radiation-related OME is usually a nonorganic disease, which is the biggest pathogenic difference between the two. However, treatment of OME following RT is still the same as that of non-radiation-related one, but the clinical efficacy is much worse than the latter. Conservative treatments such as physical and pharmacological therapy usually turn out to be ineffective. The most widely used ones are tympanocentesis and tympanostomy tube insertion. Tympanocentesis is to directly pierce the tympanic membrane and drain the middle ear effusion. However, the drainage port usually heals within 3-5 days, so it is often necessary to pierce repeatedly. The ventilation tube insertion is considered to achieve continuous drainage, but the risks of middle ear infection, slippage of ventilation tube, and permanent tympanic membrane perforation is high after the placement of tube. Therefore, the residence time of the ventilation tube is generally no more than 6-9 months.

At present, the treatments of OME following RT just deal with symptoms, instead of the cause--ETD, resulting in low cure rate, high recurrence rate and high complication rate. In recent years, balloon Eustachian tuboplasty (BET) has been performed successfully with encouraging results in patients with ETD by dilating (make larger) the cartilage segment of the Eustachian tube. However, ETD following RT used to be recognized as a contraindication to BET, possibly due to more complex pathogenesis, scruples for damage to the internal carotid artery in the lateral of the Eustachian tube, and Eustachian tube atresia. The above reasons are only speculation, and there have been already a few reports of BET being used in OME after RT for head and neck tumors.

The primary purpose of this study is to compare BET combined with tympanostomy tube insertion and simply tympanostomy tube insertion in the treatment of OME in post-radiotherapy patients on the improvement of subjective symptoms (ear fullness, etc.) and the tympanogram. The secondary purpose is to clarify the effects of BET on the incidence of middle ear infection and slippage of ventilation tube during tube retention, as well as to determine the difference of hearing improvement between the two management methods.

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed OME after radiotherapy for NPC (diagnostic criteria: have fluid drained from tympanic cavity during tympanocentesis) , who had completed radiotherapy for ≥6 months, and had failed to respond after two or more times of tympanocentesis
* Eustachian Tube Dysfunction Questionnaire score greater than 14
* clinical findings of a retracted drum
* fluid behind the drum
* tympanometry type B or C results
* patients volunteered to participate in the study and signed the informed consent
* patients volunteered to bear the corresponding costs of surgery and consumables.

Exclusion Criteria:

* NPC recurrence or other malignant tumor after radiotherapy
* a perforated tympanic membrane
* the presence of a ventilation tube
* a period of less than six months following the final radiotherapy treatment
* clear diagnosis of Eustachian ostium atresia or nasal obstruction diseases, such as severe deviated nasal septum, nasal polyp, choanal atresia, osteoradionecrosis of skull base after radiotherapy, etc.
* patients with severe underlying diseases could not tolerate general anesthesia
* patients who could not cooperate (including poor hearing and radiation encephalopathy)
* patients with other middle ear diseases, such as middle ear cholesteatoma, osteoradionecrosis of temporal bone after radiotherapy, etc.
* severe deglutition disorders
* cleft palate

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
changes in air pressure (Tympanogram) | collected at 1 month, 3 months, 6 months and 12 months after the ventilation tube removal
  Tympanogram, which measures the movement of the tympanic membrane in response to changes in air pressure, is classified by types - Type A, B and C. Each classification indicates a range that falls between normal and abnormal.

SECONDARY OUTCOMES:
Incidence of Otitis Media | 6 months post-operatively during tube retention
  The number of days of ear discharges or otorrhoea in a 6-month period of tube retention
Incidence of Slippage of Ventilation Tube | 6 months post-operatively during tube retention
  The number of times the ventilation tube falls off in a 6-month period of tube retention
Eustachian Tube Dysfunction Questionnaire (ETDQ-7) | collected at 1 month, 3 months, 6 months and 12 months after the ventilation tube removal
  The ETDQ-7 tool is used to assess the symptoms of Otitis Media With Effusion (OME), which consists of seven items with a scale of graduated responses ranging from 1 (No Problem) to 7 (Severe Problem), and 4 would correspond to a Moderate Problem. If the total score is more than 14, it is considered that there is eustachian tube dysfunction. The average post-operative ETDQ-7 score is less than 2.1 or decrease > 0.5 (minimal clinically important difference=0.5), it is considered that the eustachian tube function is improved.
Hearing gap | collected at 1 month, 3 months, 6 months and 12 months after the ventilation tube removal
  It is the change of air-bone conduction difference between pre-operation and post-operation, which is measured by Pure-Tone Audiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Xiong, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, 广东 (Guǎngdōng), China

IPD SHARING:
Plan to Share IPD: Yes